CLINICAL TRIAL: NCT03498885
Title: Preservation of the Left Colic Artery With Apical Lymph Node Dissection in Laparoscopic Rectal Cancer Surgery
Brief Title: Comparison of Low and High Ligation With Apical Lymph Node Dissection in the Laparoscopy Rectal Cancer
Acronym: PLAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: WEIDONG LIU，MD (Other)
Responsible Party: Sponsor-Investigator, WEIDONG LIU，MD, Head of Department of General Surgery, Xiangya Hospital of Central South University
Organization: Xiangya Hospital of Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCRS-1
Record Dates: First submitted 2018-01-16; First posted 2018-04-17 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; inferior mesenteric artery; Laparoscopic
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Procedure： Low ligation with apical lymph node dissection
  Procedure： High ligation with apical lymph node dissection
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low ligation (Experimental): Left colic artery (LCA) is identified, tie the sigmoid artery and superior rectal artery,Apical lymph node dissection with the left colic artery preservation is performed.
  Interventions: Procedure: Low ligation
- High ligation (Active Comparator): The IMA is ligated and divided at 2 cm from its origin. Apical lymph nodes dissection is performed.
  Interventions: Procedure: High ligation

INTERVENTIONS:
Procedure: Low ligation — Left colic artery (LCA) is identified, Tie the sigmoid artery and superior rectal artery, Apical lymph node dissection with the left colic artery preservation is performed.
  Other Names: LL
  Arms: Low ligation
Procedure: High ligation — The IMA is ligated and divided at 2 cm from its origin. Apicallymph nodes dissection is performed.
  Other Names: HL
  Arms: High ligation

SUMMARY:
The purpose of this study is to explore the different impacts of high and low ligation in laparoscopic rectal interior resection on postoperative anastomotic leakage and proximal bowel necrosis and stenosis, as well as the quality of life and long-term survival. In the anterior resection of rectum, the section level of inferior mesenteric artery (IMA) is still a controversial subject between the advocates of high and low ligation. The low ligation is defined as the IMA is ligated below the origin of the left colic artery while the high ligation refers to the IMA is ligated at its origin from the aorta. Nowadays the spread of laparoscopy has encouraged more frequent execution of the high ligation, which appears easier to achieve than the low ligation and also with the advantage of lower anastomosis traction but with the disadvantage of worse vascularization of the stumps as well.

DETAILED DESCRIPTION:
It has long been debated that whether to tie off the inferior mesenteric artery (IMA) at its origin or just below the origin of the left colic artery (LCA) of the anterior resection of the rectum. Thus far, no clear consensus has been achieved, and the level of arterial ligation still varies among institutions and patients. In the previous studies, high or low ligation takes advantage on both sides. However, there are still some researches that have demonstrated no significant difference had been found in the incidence of anastomotic leakage and other complications between the high and low ligation groups. Therefore, to provide a clear and definite answer to surgeons of how they should deal with the IMA in laparoscopy rectal surgery. We plan to explore the impacts of high and low tie in laparoscopic anterior rectal resection on postoperative anastomotic leakage and proximal bowel necrosis and stenosis, as well as the quality of life and long-term survival by prospective and multi-center clinical trial.

Surgery will be described as follows:

For low ligation group:

1. Laparoscopic surgery is performed. Tie the sigmoid artery and superior rectal artery, LCA is preserved. Lymphadenectomy to Apical lymph nodes is performed. Strip the beginning part of upper rectal artery and the first sigmoid artery. Strip the left colic artery until reaching the inferior mesenteric vein (IMV). The abdominal aorta lymph nodes need to be cleaned if it's been spotted swollen.
2. Vascular ligation level: Left colonic artery needs to be preserved, the rectal artery and the first sigmoid artery are ligated. Ligate inferior mesenteric artery below left colonic artery come across the inferior mesenteric vein level.

For high ligation groups:

Laparoscopic surgery is performed. The IMA is ligated and divided at 2 cm. from its origin. Dissect the adipose tissue and lymph nodes around IMA. The inferior mesenteric vein (IMV) is divided and ligated below the duodenal margin. The abdominal aorta lymph nodes need to be cleaned if it's been spotted swollen. For both groups Total Mesolectal Excision (TME) is performed according to the principles of Heald.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 75 Years (Adult, Senior).
* Colonoscopy and pathology shows rectal or sigmoid adenocarcinoma.
* Tumor located at 4-15 cm from the dentate line.
* The clinical staging of tumor by MRI within T1-4a when tumor Above the peritoneum and T3N0-2 when tumor below the peritoneum.
* Receive or not receive neoadjuvant chemotherapy based on 5-fluorouracil before surgery and radical resection is available after neoadjuvant chemotherapy.
* Anus-saving operation is available.
* ASA class: I-III.
* Well tolerate to general anesthesia.
* ECOG score: 0-1.
* Patients - can understand and are willing to take part in the clinical trial.

Exclusion Criteria:

* Severe cardiovascular disease, uncontrollable infection or other severe complications.
* Severe mental illness.
* Suffer with other carcinoma simultaneously or sequentially in 5 years.
* Familial polyposis coli or Multiple -colorectal tumor.
* History of abdominal surgery and with severe abdominal adhesions.
* Combine with acute intestinal obstruction, intestinal bleeding, intestinal perforation and emergency surgery is needed.
* Multiple organs resection surgery is needed.
* Abdominoperineal resection need to be performed.
* ASA class: IV to V.
* Pregnant, suckling period or reject to birth control.
* Patient who unable to go through the clinical trial because of familial,social or religious factors.
* Refuse to take part in the trial.
* Patients without an informed consent.
* Non-compliant patient
* The patient or their family members want to withdraw from the clinical trial.
* Loss to follow-up
* Researchers think the participants need to withdraw from the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage | 3 months
  Anastomosis leakage rate after surgery, acute or chronic

SECONDARY OUTCOMES:
proximal bowel necrosis | 3 months
  Proximal bowel necrosis rate after surgery, acute or chronic
proximal bowel stenosis | 3 months
  Proximal bowel stenosis rate after surgery, acute or chronic
Characteristics of the division branches of the inferior mesenteric artery in Chinese people | 1-2 days
  e.g.,The distance from the left colon artery to the root of inferior mesenteric artery(cm).
Apical Lymph Nodes Positive Rate | 14 days
  Apical Lymph Nodes Positive Rate
Conversion rate to laparotomy | 5-years
  Conversion rate to laparotomy
Complications of defunctioning stoma | 3 months
  Complications of defunctioning stoma
Early postoperative complications: Anastomotic bleeding, etc. | 30 days
  Early postoperative complications: Anastomotic bleeding, etc.
Anastomosis stenosis rate after surgery | 30 days
  Anastomosis stenosis rate after surgery
Mortality rate in 3 months after surgery | 3 months
  Mortality rate in 3 months after surgery
Life quality | 5-years
  Life quality is measured by questionnaire(EORTC QLQ-C30 (version 3)).
Micturition function scoring | 3 months
  Micturition function is measured by questionnaire(IPSS).
Sexual function scoring | 3 months
  Sexual function is measured by questionnaire(The IIEF-5 questionnaire).
5-years overall survival rate | 5-years
  5-years overall survival rate
5-years disease free survival rate | 5-years
  5-years disease free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Wei dong Liu, MD, Principal Investigator — Xiangya Hospital of Central South University; Xi Xie, MD, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
we would like to share our data.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Around 2025
Access Criteria: Someone who has the same or similar research could contact us at davidcsu@foxmail.com

REFERENCES:
- [Background] Milnerowicz S, Milnerowicz A, Tabola R. A middle mesenteric artery. Surg Radiol Anat. 2012 Dec;34(10):973-5. doi: 10.1007/s00276-012-0987-y. Epub 2012 Jul 22. PMID 22820922
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Kim DI, Han SH. A rare branching pattern of hindgut: absence of inferior mesenteric artery. Surg Radiol Anat. 2017 Jul;39(7):803-806. doi: 10.1007/s00276-016-1770-2. Epub 2016 Dec 20. PMID 27999945
- [Background] Vermeer TA, Orsini RG, Daams F, Nieuwenhuijzen GA, Rutten HJ. Anastomotic leakage and presacral abscess formation after locally advanced rectal cancer surgery: Incidence, risk factors and treatment. Eur J Surg Oncol. 2014 Nov;40(11):1502-9. doi: 10.1016/j.ejso.2014.03.019. Epub 2014 Apr 4. PMID 24745995
- [Background] Abe T, Ujiie A, Taguchi Y, Satoh S, Shibuya T, Jun Y, Isogai S, Satoh YI. Anomalous inferior mesenteric artery supplying the ascending, transverse, descending, and sigmoid colons. Anat Sci Int. 2018 Jan;93(1):144-148. doi: 10.1007/s12565-017-0401-2. Epub 2017 Apr 6. PMID 28386743
- [Background] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450
- [Background] Smedh K, Sverrisson I, Chabok A, Nikberg M; HAPIrect Collaborative Study Group. Hartmann's procedure vs abdominoperineal resection with intersphincteric dissection in patients with rectal cancer: a randomized multicentre trial (HAPIrect). BMC Surg. 2016 Jul 11;16(1):43. doi: 10.1186/s12893-016-0161-2. PMID 27401339
- [Background] Hida J, Yasutomi M, Maruyama T, Uchida T, Nakajima A, Wakano T, Tokoro T, Kubo R. High ligation of the inferior mesenteric artery with hypogastric nerve preservation in rectal cancer surgery. Surg Today. 1999;29(5):482-3. doi: 10.1007/BF02483047. PMID 10333426
- [Background] Mari G, Maggioni D, Costanzi A, Miranda A, Rigamonti L, Crippa J, Magistro C, Di Lernia S, Forgione A, Carnevali P, Nichelatti M, Carzaniga P, Valenti F, Rovagnati M, Berselli M, Cocozza E, Livraghi L, Origi M, Scandroglio I, Roscio F, De Luca A, Ferrari G, Pugliese R. "High or low Inferior Mesenteric Artery ligation in Laparoscopic low Anterior Resection: study protocol for a randomized controlled trial" (HIGHLOW trial). Trials. 2015 Jan 27;16:21. doi: 10.1186/s13063-014-0537-5. PMID 25623323
- [Background] Titu LV, Tweedle E, Rooney PS. High tie of the inferior mesenteric artery in curative surgery for left colonic and rectal cancers: a systematic review. Dig Surg. 2008;25(2):148-57. doi: 10.1159/000128172. Epub 2008 Apr 29. PMID 18446037
- [Background] Hall NR, Finan PJ, Stephenson BM, Lowndes RH, Young HL. High tie of the inferior mesenteric artery in distal colorectal resections--a safe vascular procedure. Int J Colorectal Dis. 1995;10(1):29-32. doi: 10.1007/BF00337583. PMID 7745320
- [Background] Cirocchi R, Farinella E, Trastulli S, Desiderio J, Di Rocco G, Covarelli P, Santoro A, Giustozzi G, Redler A, Avenia N, Rulli A, Noya G, Boselli C. High tie versus low tie of the inferior mesenteric artery: a protocol for a systematic review. World J Surg Oncol. 2011 Nov 9;9:147. doi: 10.1186/1477-7819-9-147. PMID 22071020
- [Background] Bertrand MM, Delmond L, Mazars R, Ripoche J, Macri F, Prudhomme M. Is low tie ligation truly reproducible in colorectal cancer surgery? Anatomical study of the inferior mesenteric artery division branches. Surg Radiol Anat. 2014 Dec;36(10):1057-62. doi: 10.1007/s00276-014-1281-y. Epub 2014 Mar 15. PMID 24633578
- [Background] BERNSTEIN WC, BERNSTEIN EF. Ischemic ulcerative colitis following inferior mesenteric arterial ligation. Dis Colon Rectum. 1963 Jan-Feb;6:54-61. doi: 10.1007/BF02617232. No abstract available. PMID 13967713
- [Background] Francone E, Bonfante P, Bruno MS, Intersimone D, Falco E, Berti S. Laparoscopic Inferior Mesenteric Artery Peeling: An Alternative to High or Low Vascular Ligation for Sigmoid Colon Cancer Resection. World J Surg. 2016 Nov;40(11):2790-2795. doi: 10.1007/s00268-016-3611-1. PMID 27334448
- [Background] Zhang W, Lou Z, Liu Q, Meng R, Gong H, Hao L, Liu P, Sun G, Ma J, Zhang W. Multicenter analysis of risk factors for anastomotic leakage after middle and low rectal cancer resection without diverting stoma: a retrospective study of 319 consecutive patients. Int J Colorectal Dis. 2017 Oct;32(10):1431-1437. doi: 10.1007/s00384-017-2875-8. Epub 2017 Aug 2. PMID 28766076
- [Background] Miyamoto R, Nagai K, Kemmochi A, Inagawa S, Yamamoto M. Three-dimensional reconstruction of the vascular arrangement including the inferior mesenteric artery and left colic artery in laparoscope-assisted colorectal surgery. Surg Endosc. 2016 Oct;30(10):4400-4. doi: 10.1007/s00464-016-4758-4. Epub 2016 Feb 5. PMID 26850027
- [Background] Michelson H, Bolund C, Nilsson B, Brandberg Y. Health-related quality of life measured by the EORTC QLQ-C30--reference values from a large sample of Swedish population. Acta Oncol. 2000;39(4):477-84. doi: 10.1080/028418600750013384. PMID 11041109
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Background] Rosen RC, Cappelleri JC, Smith MD, Lipsky J, Pena BM. Development and evaluation of an abridged, 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool for erectile dysfunction. Int J Impot Res. 1999 Dec;11(6):319-26. doi: 10.1038/sj.ijir.3900472. PMID 10637462